CLINICAL TRIAL: NCT03855904
Title: The Efficacy of Hemostatic Powder TC-325 Versus Standard Endoscopic Treatment for Gastrointestinal Bleeding From Malignancy; a Multi-center Randomized Trial
Brief Title: HemosprayTM for Gastrointestinal Bleeding From Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Principle investigator, Gastrointestinal Unit, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RP014
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Gastrointestinal Bleeding From Malignancy
Keywords: GI bleeding; Hemospray; TC-325; malignancy; tumor
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Neoplasms

STUDY DESIGN:
Intervention Model Description: At the time of initial early endoscopy, following fulfillment of patient and bleeding lesion eligibility, central randomization is carried out in a 1:1 ratio, in blocks of 4. The confidential centralized random numbers allocation is obtained by using REDCap (https://www.project-redcap.org/), a web based platform available to all participating centres. An independent staff member maintained the randomization numbers in sealed opaque envelopes. After obtaining a written informed from an eligible patient, the gastroenterologists who were blinded to the sequence of treatment opened the next numbered sealed envelope with treatment allocation.Randomization is stratified by location of bleed (upper versus lower GI tract), considering the lack of comparative outcomes data in the literature, thus balancing known and unknown confounding more completely
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention and control arms, blinding of the endoscopist is not possible (visual clues as to the nature of endoscopic treatment are evident and no sham procedure can be delivered since both are active treatment groups). However, in order to minimize possible patient/observer bias, any research team member or investigator assessing the patient after the initial endoscopy and involved in data collection or analysis, as well as the patient, and research nurse will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TC-325 (Experimental): The intervention (experimental) arm patients are treated initially with TC-325 alone. Treatment failure for TC-325 is defined as endoscopists cannot achieve hemostasis with 1 syringe (20gm) of TC-325.
  Interventions: Device: TC-325
- Traditional treatment (Control group) (Active Comparator): Control group patients initially receive usual standard of (traditional) endoscopic treatment (SET) as defined by injection therapy with another modality or sole/combination use of thermal or mechanical modalities. Crossovers to either treatment arm are permitted if immediate haemostasis does not achieved with standard endoscopic or TC-325 application.Treatment failure of SET is defined as endoscopists cannot achieve hemostasis by selected SET.
  Interventions: Device: TC-325

INTERVENTIONS:
Device: TC-325 — TC-325 compounds of inorganic, non-absorbable powder which acts locally at the mucosal tissue. When spraying the powder on to the blood, it will become a stable barrier sheet because of the effect of clotting factors accumulation and, then the normal healing process can be promoted.
  Other Names: HemosprayTM

SUMMARY:
Title: The efficacy of hemostatic powder TC-325 versus standard endoscopic treatment for gastrointestinal bleeding from malignancy; a multi-center randomized trial

Background: Gastrointestinal (GI) bleeding arising from malignant tumors is increasingly recognized as a result of oncological advances and improved detection methods. However, conventional endoscopic hemostatic methods are not reliable to control bleeding. It has a trend to be an effective hemostasis method for active GI bleeding from tumor, however, in view of the lack of RCTs and large-scale studies, the efficacy of TC-325 is still inconclusive.

Objective: To evaluate the efficacy of TC325 in endoscopic hemostasis treatment for malignant gastrointestinal hemorrhage.The 24-hour, 72-hour, 30-day, 90-day and 180-day rebleeding rate were assessed as the outcomes of treatment as well as 6-month mortality.

Study design: Single-blinded, multi-center, randomized-control trial study The intervention (experimental) arm: TC-325 alone (define failure if continued bleeding despite application of 1 syringes) The control arm: Standard of (traditional) endoscopic treatments

** Crossover is possible. Inclusion criteria: Patients with acute upper or lower GIB from a lesion that is actively bleeding at index endoscopy (spurting or oozing) and is suspected to be malignant or diagnosed as malignancy from previous tissue diagnosis.

Exclusion criteria: Patients less than 18 years old, previously included in the trial, ECOG score 3 or 4, pregnancy/lactation, and/or bleeding from GI sources suspected of not being malignant. If an endoscopist is unsure of the malignant likelihood of the lesion, he/she will not be enrolled.

Sample size: 112 in total

Duration of participation for each volunteer: 180 days

ELIGIBILITY:
Inclusion Criteria:

* Acute upper or lower gastrointestinal bleeding
* Endoscopy shows actively bleeding at index endoscopy (spurting or oozing)
* Bleeding from malignancy

Exclusion Criteria:

* Less than 18 years old
* Previously included in the trial
* Eastern Cooperative Oncology Group (ECOG) score 3 or 4
* Pregnancy/lactation
* Bleeding from GI sources suspected of not being malignant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of TC-325 in preventing 30-day rebleeding following the index malignant hemorrhage: Rebleeding rate | 30 days
  Rebleeding rate

SECONDARY OUTCOMES:
1. To evaluate the efficacy of TC-325 in immediate hemostasis and rebleeding at 24 hours, 72 hours, 90 days and 180 days following presentation at initial bleeding episode as well as 6-month survival rate | 180 days
  Morbidity and mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Rapat Pittayanon, MD, Principal Investigator — King Chulalongkorn Memorial Hospital
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data to others.

REFERENCES:
- [Derived] Pittayanon R, Khongka W, Linlawan S, Thungsuk R, Aumkaew S, Teeratorn N, Maytapa J, Kimtrakool S, Pakvisal P, Kongtub N, Rerknimitr R, Barkun A. Hemostatic Powder vs Standard Endoscopic Treatment for Gastrointestinal Tumor Bleeding: A Multicenter Randomized Trial. Gastroenterology. 2023 Sep;165(3):762-772.e2. doi: 10.1053/j.gastro.2023.05.042. Epub 2023 Jun 3. PMID 37277078